CLINICAL TRIAL: NCT03683329
Title: Antibiotic De-escalation in Onco-hematology Patients for Sepsis or Septic Shock
Acronym: DéPOH
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Institut Paoli-Calmettes (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: DéPOH-IPC 2015-022
Record Dates: First submitted 2018-08-12; First posted 2018-09-25 (Actual); Last update posted 2026-01-22 (Actual); Status verified 2025-04

CONDITIONS: Critical Care; Cancer
Keywords: critical care; cancer; antimicrobial treatment; de-escalation; septic shock; sepsis
MeSH Terms: conditions — Neoplasms; Shock, Septic; Sepsis

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Antibiotic de-escalation (Experimental): * According to the results of the antibiogram of the suspected causative bacteria, the ''pivotal'' antibiotic (antipseudomonal betalactam) used for empirical treatment is switched to an antibiotic with a spectrum as narrow as possible according to the targeted pathogens,
  * Stop the companion antibiotic (aminoglycoside, fluoroquinolone, macrolide) between day 2 and day 3 of antibiotic treatment as much as possible,
  * Stop the empirical antibiotic directed against methicillin-resistant staphylococcus aureus (MRSA) or an enterococcus in the absence of these bacteria in the culture.
  Interventions: Other: Antibiotic de-escalation
- Standard treatment without de-escalation (Active Comparator): * The companion antibiotic is stopped between day 3 and day 5 of antibiotic treatment as much as possible and according to the local prescription,
  * Empirical antibiotics directed against MRSA or enterococcus were used according to local prescription and/or international guidelines,
  * The pivotal antibiotic of the empirical treatment is continued for the entire duration of the treatment, independently of microbiological results. For prolonged treatment, the physician has the choice of de-escalating after 8-15 days of treatment.
  Interventions: Other: Standard treatment

INTERVENTIONS:
Other: Antibiotic de-escalation — All the therapeutic protocols made the object of a consensus between the different partners of the study.
  Antibiotic treatment will be delivered according to current practice, in agreement with the national and international recommendation.
  Arms: Antibiotic de-escalation
Other: Standard treatment — Antibiotic treatment will be delivered according to current practice, in agreement with the national and international recommendation.
  Arms: Standard treatment without de-escalation

SUMMARY:
De-escalation aims at reducing the use of broad-spectrum antibiotics and therefore the emergence of multidrug-resistant (MDR) pathogens.

Observational studies suggested that this strategy seems to be safe. However, there is no adequate, direct evidence showing de-escalation of antimicrobial agents to be effective and safe for onco-hematology patients with sepsis or septic shock. Thus, randomized clinical trials are needed for testing the safety and efficiency of de-escalation of antimicrobial therapy.

The investigator's hypothesis is that de-escalation of empirical antimicrobial therapy in onco-hematology patients with sepsis or septic shock is noninferior to the continuation of empirical antimicrobial therapy.

The first aim of the study is to demonstrate that de-escalation is noninferior to the continuation of broad-spectrum antibiotics in terms of hospital mortality.

The secondary aims are to compare the two strategies in terms of mortality, duration of antimicrobial therapy, durations of mechanical ventilation, vasopressor use, numbers of superinfections, organ failure.

Antimicrobial de-escalation (ADE) of antimicrobial therapy is a strategy proposed to allow for the rational use of broad-spectrum antimicrobial therapy as the empiric treatment for infections and minimize the overall exposure to these broad-spectrum agents. The need for prompt, effective antimicrobial therapy for patients with known or suspected infections is widely accepted. This principle leads to the use of very broad-spectrum antimicrobial therapy to increase the odds that all suspected potential pathogens are adequately treated. However, the potential drawback is selection of multidrug-resistant (MDR) organisms.

ADE is widely recommended in the management of antimicrobial therapy in intensive care unit (ICU) patients. The Surviving Sepsis Campaign guidelines describe and recommend the process for selecting antimicrobial therapy as commencement of antimicrobials within the first hour, antimicrobial therapy broad enough to cover all likely pathogens, and daily reassessment for potential ADE.

To date, no randomized study assessing this strategy is available for this specific population of cancer critically ill patients. In a recent systematic review based on 13 observational studies and one randomized controlled trial, the authors conclude that the equipoise remains and a large randomized trial is required to assess the effect of the antibiotics de-escalation strategy on the bacterial ecosystem, on MDR carriage, and on patient outcomes.

DETAILED DESCRIPTION:
An interim analysis planned after inclusion of 233 patients.

* Subgroup analyses will be performed on patient subsets:

* Patients with allogeneic hematopoietic stem cell transplant,
* Neutropenic patients (Neutrophils < 0.5 Giga/L),
* Hematological disease,
* Oncological disease,
* Polymicrobial sepsis,
* Multi-drug resistant organisms,
* Patients presenting with bacterial pneumoniae,
* Patients presenting with Intra-abdominal infection,
* Patients presenting with bacteraemia,
* Patients presenting with gram negative bacteria infection,
* Patients presenting with gram positive cocci infection,
* Patients presenting with septic shock,
* Patients presenting with sepsis.

ELIGIBILITY:
Inclusion Criteria:

1. Written informed consent from the patient or proxy (if present) before inclusion or once possible when patient has been included in a context of emergency
2. Age ≥ 18 years,
3. Onco-hematology patient admitted to intensive care for sepsis or septic shock according to the following criteria:

   * Sepsis:

     * A suspected infection
     * And an acute increase of ≥ 2 SOFA points (a proxy for organ dysfunction)
   * Septic shock:

     * sepsis
     * and vasopressor therapy needed to elevate MAP ≥65 mm Hg and lactate >2 mmol/L despite adequate fluid resuscitation
4. Patient treated with an empirical antibiotic treatment,
5. Patient with at least one microbiological sample collected at least within the first 48 hours following the diagnosis of sepsis in ICU
6. Patient with an identified infectious site according to the definitions,
7. Patient with an identified bacteria microorganism after microbiological examination,
8. Patient affiliated to the national French statutory healthcare insurance system or beneficiary of this regimen.

Exclusion Criteria:

1. Patient colonized with a multi-drug resistant organisms preventing de-escalation antibiotic,
2. Pregnant or breast-feeding woman,
3. No affiliation to the national French statutory healthcare insurance system,
4. Patients deprived of liberty or placed under the authority of a tutor,
5. Inappropriate probabilistic antibiotic treatment,
6. Expected mortality within 48 hours,
7. Patient admitted to the ICU for end-of-life care (do-not-resuscitate patients) . Do-not-intubate (DNI) patients can be included.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 368 (Actual)
Dates: Start 2018-11-26 (Actual); Primary Completion 2024-07-26 (Actual); Study Completion 2024-07-26 (Actual)

PRIMARY OUTCOMES:
Hospital mortality | From day of inclusion until day of ICU discharge, up to 3 months
  death from any cause during hospital stay

SECONDARY OUTCOMES:
Death | From day of inclusion until ICU discharge, day 28 and day 90
  death from any cause into the ICU, day 28 and day 90
ICU length of stay | From day of inclusion until ICU discharge (until day 90)
Hospital length of stay | From day of inclusion until ICU discharge (until day 90)
Severe organ dysfunctions | From day of inclusion until ICU discharge (until day 90)
  A Sepsis-related Organ Failure Assessment (SOFA) score>2 for each organ (respiratory, hematologic, cardiac, neurologic, hepatic, renal)
Respiratory dysfunction-free days at day 28 | from inclusion to day 28
  days without respiratory dysfunction (respiratory SOFA score<3)
Renal dysfunction-free days at day 28 | from inclusion to day 28
  days without renal dysfunction (renal SOFA score<3)
Neurologic dysfunction-free days at day 28 | from inclusion to day 28
  days without neurologic dysfunction (neurologic SOFA score<3)
Cardiac dysfunction-free days at day 28 | from inclusion to day 28
  days without cardiac dysfunction (cardiac SOFA score<3)
Hepatic dysfunction-free days at day 28 | From inclusion to day 28
  days without hepatic dysfunction (hepatic SOFA score<3)
Hematologic dysfunction-free days at day 28 | From inclusion to day 28
  days without hematologic dysfunction (hematologic SOFA score<3)
Ventilator-free days at day 28 | From inclusion to day 28
  days without invasive mechanical ventilation
Vasopressors-free days at day 28 | From inclusion to day 28
  days without vasopressors treatment
Dialysis-free days at day 28 | From inclusion to day 28
  days without dialysis treatment
Duration of antibiotic treatment during ICU stay | From day of admission to ICU until day 90
  Duration between the first antibiotic initiation and the last antibiotic stop
Number of antibiotics de-escalated | From inclusion to ICU discharge until day 90
  Number of antibiotics de-escalated in each arm
Number of antifungal de-escalated | From inclusion to ICU discharge until day 90
  Number of antifungal de-escalated in each arm
Number of antiviral de-escalated | From inclusion to ICU discharge until day 90
  Number of antiviral de-escalated in each arm
Antibiotic-free days at day 28 | From inclusion to day 28
  days without antibiotic treatment
Antibiotic-free days during ICU stay | From admission to ICU to ICU discharge until day 90
  days without antibiotic treatment
Antibiotic-free days during hospital stay | From admission to ICU to hospital discharge until day 90
  Days without antibiotic treatment
Antibiotic-free days at day 90 | From admission to ICU to day 90
  Days without antibiotic treatment
Antifungal-free days at day 28 | From admission to ICU to day 28
  Days without antifungal treatment
Antiviral-free days at day 28 | From admission to ICU to day 28
  Days without antiviral treatment
Antifungal-free days during ICU stay | From admission to ICU to ICU discharge until day 90
  Days without antifungal treatment
Antiviral-free days during ICU stay | From admission to ICU to ICU discharge until day 90
  Days without antiviral treatment
Antiviral-free days during hospital stay | From admission to ICU to hospital discharge until day 90
  Days without antiviral treatment
Antifungal-free days during hospital stay | From admission to ICU to hospital discharge until day 90
  Days without antifungal treatment
Antifungal-free days at day 90 | From admission to ICU to day 90
  Days without antifungal treatment
Antiviral-free days at day 90 | From admission to ICU to day 90
  Days without antiviral treatment
Number of days of exposure to each antibiotic per 1000 inpatient days | From admission to ICU to ICU discharge until day 90
  For the entire cohort:(number of antibiotic days / number of ICU days)*1000
Number of days of exposure to each antifungal per 1000 inpatient days | From admission to ICU to ICU discharge until day 90
  For the entire cohort:(number of antifungal days / number of ICU days)*1000
Number of days of exposure to each antiviral per 1000 inpatient days | From admission to ICU to ICU discharge until day 90
  For the entire cohort:(number of antiviral days / number of ICU days)*1000
Adverse events | From inclusion to ICU discharge until day 90
  Adverse events assessed according to the Common Toxicity Criteria for Adverse Events (CTCAE) version 5.0
Compliance to de-escalation strategy | From inclusion to ICU discharge until day 90
  number of patients de-escalated/number of patients included in the experimental arm
Compliance to the continuation strategy | From inclusion to ICU discharge until day 90
  number of patients not de-escalated/number of patients included in the continuation group
Percentage of emerging multidrug-resistant bacteria | From inclusion until day 28
  Percentage of emerging multidrug-resistant bacteria isolated from specimen taken for routine microbiological assessments
Cost of antibiotic treatment | From inclusion to ICU discharge until day 90
Patients presenting with bacterial pneumoniae, | From inclusion to ICU discharge until day 90
Patients presenting with Intra-abdominal infection. | From inclusion to ICU discharge until day 90
Patients presenting with bacteraemia | From inclusion to ICU discharge until day 90
Number of patients in the de-escalation group without de-escalation | From inclusion to ICU discharge until day 90
Rate of new infectious episode requiring a new antibiotic treatment | From inclusion to ICU discharge until day 90
Rate of patients requiring an escalation after de-escalation | From inclusion to ICU discharge until day 90
Rate of recovery from infection | From inclusion to ICU discharge until day 90

CONTACTS AND LOCATIONS:
Overall Officials: MOKART Djamel, MD, Principal Investigator — Institut Paoli-Calmettes
Locations (1):
- Institut Paoli Calmettes, Marseille, France

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- See also: Institut Paoli-Calmettes — http://institutpaolicalmettes.fr